CLINICAL TRIAL: NCT01722071
Title: Deciphering the Role of Oxytocin in Motivation: an fMRI Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tiffany Love (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Tiffany Love, Research Investigator, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UL1RR024986 (NIH)
Record Dates: First submitted 2012-10-29; First posted 2012-11-06 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Focus of Study: Neural Correlates of Oxytocin Administration
Keywords: Oxytocin; Functional Magnetic Resonance Imaging; Social; Motivation
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Each participant will be studied using fMRI following self-administration of placebo.
  Interventions: Drug: Placebo
- Oxytocin (Experimental): Each participant will be studied using fMRI following self-administration of oxytocin.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Placebo — Placebo intranasal administration, 3 puffs per nostril delivered approximately 30 minutes prior to scanning session.
  Arms: Placebo
Drug: Oxytocin — Oxytocin intranasal administration, 24 IU, 3 puffs per nostril at 4 IU per puff delivered approximately 30 minutes prior to scanning session.
  Other Names: Syntocinon®
  Arms: Oxytocin

SUMMARY:
The proposed study will investigate the effects of intranasal oxytocin administration on neural activity associated with social and non-social motivation.

DETAILED DESCRIPTION:
Oxytocin is a well-known social and reproductive hormone demonstrated to have a variety of prosocial effects in humans including enhancing trust and generosity, improving positive communication, increasing eye gaze, and reducing anxiety. Oxytocin is hypothesized to facilitate social behaviors via its modulation of motivational networks. With this study, we will characterize oxytocin's effects on the neural processing of salient stimuli. We will utilize a noninvasive brain imaging technique, functional magnetic resonance imaging (fMRI), to assess brain activity while participants perform tests designed to engage neural circuits associated with the processing of social and non-social stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 20-35 years of age at the time of screening
* Right-handedness
* Non-smoking
* No current or past history of neurological or psychiatric illness, including substance abuse or dependence
* No acute medical illness
* Written informed consent obtained from subject

Exclusion Criteria:

* Female
* Left-handedness or ambidextrous
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Known allergies to oxytocin or to preservatives in the nasal spray
* Participants who exhibit nasal obstruction or upper-respiratory tract infection at the time of scanning or report the use of intranasally administered medications for up to two weeks prior to screening
* Participants unable to tolerate the scanning procedures or would be unfit for scanning purposes (e.g. metal implants, claustrophobic, unable to lie still for the duration of the scan)
* Any current or past history of medical, neurological, or psychiatric illness or family history of psychiatric or neurologic disease in first-degree relatives
* Neurological illness, abnormal MRI (except if due to technical factors)
* Acute or uncorrected medical illnesses, including history of hepatic or renal dysfunction.
* Participants currently taking medications including any treatment, current or past with antipsychotics, mood stabilizers, isoniazid, glucocorticoids, psychostimulants and psychostimulant appetite suppressants, or centrally active antihypertensive drugs (e.g., clonidine, reserpine).
* Treatment within six months with any of the following: hormone use (testosterone, DHEA), antidepressants, opioid drugs.
* Treatment within one month with sedative hypnotic medications (benzodiazepines, barbiturates), or over the counter sleeping aids
* Current or past history of substance abuse or dependence
* Any reported lifetime use of any category of illicit drugs
* Positive urine drug screen

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany M Love, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Mickey BJ, Heffernan J, Heisel C, Pecina M, Hsu DT, Zubieta JK, Love TM. Oxytocin modulates hemodynamic responses to monetary incentives in humans. Psychopharmacology (Berl). 2016 Dec;233(23-24):3905-3919. doi: 10.1007/s00213-016-4423-6. Epub 2016 Sep 10. PMID 27614896

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Oxytocin: These participants were first studied using fMRI following self-administration of placebo (followed by another scanning session with oxytocin).
  Placebo: Placebo intranasal administration, 3 puffs per nostril delivered approximately 30 minutes prior to scanning session.
- Oxytocin Then Placebo: These participants were first studied using fMRI following self-administration of oxytocin (followed by another scanning session with placebo).
  Oxytocin: Oxytocin intranasal administration, 24 IU, 3 puffs per nostril at 4 IU per puff delivered approximately 30 minutes prior to scanning session.
Period: Overall Study
Arm/Group | Placebo Then Oxytocin | Oxytocin Then Placebo
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who completed Baseline Assessments prior to scanning.
Groups:
- Participants: Each participant will complete baseline assessments prior to being studied using fMRI
Arm/Group | Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Data: Change in BOLD Activity Between Placebo and Oxytocin Treatment.
Description: Drug effect will be assessed by ascertaining changes in brain activity between placebo and oxytocin sessions.
  Imaging data will be analyzed from all subjects in a final analysis. Individual subject analyses will be done on a bimonthly basis.
  Results represent neural responses to the anticipation of an uncertain reward within the Nucleus Accumbens (Bilateral). These are given as beta values (i.e. parameter estimates).
Time Frame: Change from Week 1, Day 1 (Scan 1) and Scan 2 (within the first 30 days after scan 1).
Population: Only 8 participants' BOLD data were included in the final group analysis in the Placebo then Oxytocin arm -- 1 participant was excluded from the study prior to scanning, 1 participant was scanned but due to technical issues the BOLD data was not used.
Measure: Mean (Standard Error); unit: BOLD signal change (beta values)
Groups:
- Placebo Then Oxytocin: Each participant will be studied using fMRI following self-administration of placebo.
  Placebo: Placebo intranasal administration, 3 puffs per nostril delivered approximately 30 minutes prior to scanning session.
- Oxytocin Then Placebo: Each participant will be studied using fMRI following self-administration of oxytocin.
  Oxytocin: Oxytocin intranasal administration, 24 IU, 3 puffs per nostril at 4 IU per puff delivered approximately 30 minutes prior to scanning session.
Arm/Group | Placebo Then Oxytocin | Oxytocin Then Placebo
Number analyzed (Participants) | 8 | 10
BOLD signal change (beta values)
  Placebo | 0.7944 (0.3252) | 0.5790 (0.2515)
  Oxytocin | 0.6119 (0.2040) | 0.6688 (0.3642)
Statistical Analysis 1: Comparison: Placebo Then Oxytocin vs Oxytocin Then Placebo; A two-sided paired t-test was performed to determine whether oxytocin administration was associated with reward-related BOLD signal changes (within the Nucleus Accumbens [Bilateral]). For the group of 18 participants, BOLD signal activity was compared between oxytocin and placebo scanning days; Test type: Superiority or Other; p = 0.890, t-test, 2 sided — The a priori threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: Placebo Then Oxytocin; A two-sided paired t-test was performed to determine whether oxytocin administration was associated with reward-related BOLD signal changes (within the Nucleus Accumbens [Bilateral]). For the group of 8 participants, BOLD signal activity was compared between oxytocin and placebo scanning days; Test type: Superiority or Other; p = 0.422, t-test, 2 sided — The a priori threshold for statistical significance was p<0.05
Statistical Analysis 3: Comparison: Oxytocin Then Placebo; A two-sided paired t-test was performed to determine whether oxytocin administration was associated with reward-related BOLD signal changes (within the Nucleus Accumbens [Bilateral]). For the group of 10 participants, BOLD signal activity was compared between oxytocin and placebo scanning days; Test type: Superiority or Other; p = 0.814, t-test, 2 sided — The a priori threshold for statistical significance was p<0.05

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on each scanning day and 24 hours later (i.e. assessed at 4 different time points for each participant).
Description: Serious adverse events were collected/assessed, but none were observed.
Arm/Group | Placebo Then Oxytocin | Oxytocin Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes